CLINICAL TRIAL: NCT00496353
Title: A Phase I/II Dose Escalation and Proof-of-Concept Study of MK2461 in Patients With Advanced Solid Tumors
Brief Title: MK2461 Phase I/II Study in Patients With Advanced Solid Tumors (MK-2461-002 AM1)(COMPLETED)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2461-002; 2007_016
Record Dates: First submitted 2007-07-02; First posted 2007-07-04 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Neoplasm
Keywords: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms | interventions — 5H-benzo(4,5)cyclohepta(1,2-b)pyridin-5-one

INTERVENTIONS:
Drug: MK2461 — MK2461 treatment, bid, 28-day

SUMMARY:
The purposes of this phase I portion are; 1) to evaluate the safety and tolerability of MK2461 and 2) to determine the recommended phase 2 dose or doses of MK2461.

The purpose of the phase II portion is to evaluate the anti-tumor efficacy of MK2461.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age, with adequate organ function, and an ecog performance of <2

Exclusion Criteria:

* No chemotherapy, radiotherapy, or biological therapy with 4 weeks of study participation
* Patients must not have primary central nervous system tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-06; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of MK2461 by assessing incidence of toxicities. Pharmacokinetic and pharmacodynamic parameter will be evaluated. | 18 Months

SECONDARY OUTCOMES:
To evaluate the anti-tumor efficacy of MK2461 in patients with advanced solid tumor by assessing the response rate, progression- free survival, duration of response, time to response and time to progression. | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC